CLINICAL TRIAL: NCT01326052
Title: Effect of Inferior Mesenteric Artery Preservation Performing Left Hemicolectomy for Diverticulosis in the Anorectal Function
Brief Title: Improvement of Anorectal Function While Preserving of Inferior Mesenteric Artery Performing Left Hemicolectomy for Diverticulosis
Acronym: IPIMAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, Reserch Fellows, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS-004
Record Dates: First submitted 2011-03-25; First posted 2011-03-30 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Defecatory Disorders After Left Colonic or Rectal Resection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inferior Mesenteric Artery Preservation (Experimental): Performing left hemicolectomy the IMA was preserved ligating close to the colonic wall the sigmoids arteries.
  Interventions: Procedure: Inferior Mesenteric Artery Preservation
- Inferior Mesenteric Artery Ligation (Active Comparator): Performing left hemicolectomy the IMA is ligated and sectioned after the origin of left colic artery
  Interventions: Procedure: Inferior Mesenteric Artery Ligation

INTERVENTIONS:
Procedure: Inferior Mesenteric Artery Preservation — Performing left hemicolectomy the IMA was preserved ligating close to the colonic wall the sigmoids arteries.
  Other Names: IMA-P
  Arms: Inferior Mesenteric Artery Preservation
Procedure: Inferior Mesenteric Artery Ligation — Performing left hemicolectomy the IMA is ligated and sectioned after the origin of left colic artery
  Other Names: IMA-L
  Arms: Inferior Mesenteric Artery Ligation

SUMMARY:
The aim of the study is to evaluate the anorectal function after hemicolectomy if we preserve or not the Inferior Mesenteric Artery (IMA). This study wants to demonstrate that IMA preservation could improve patient's quality of life reducing incontinence and/or constipation rate.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 80 years
* BMI<35
* Presence of symptomatic diverticular disease
* ASA I-III

Exclusion Criteria:

* age > 80 years
* BMI>35
* ASA IV
* Hinchey III-IV
* Past performed procedure that could be modify the nervous pattern (i.e. colorectal surgery, left nephrectomy, hysteroannessectomy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-01; Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from preoperative time in anorectal function | 6 and 12 months
  We evaluate the presence of modification in anorectal function respect to the preoperative time. This is assessed with specific questionnnaires and anorectal manometry

SECONDARY OUTCOMES:
Constipation | 6 and 12 months
  We evaluate with a questionnaire (Constipation scoring system) the presence of postoperative constipation
Incontinence | 6 and 12 months
  We evaluate with a questionnaire (Continence scale), anorectal manometry and eventually with endoanal ultrasonography the precence of incontinence
Quality of life | 6 and 12 months
  We evaluate with SF-36 questionnaire the postoperative quality of life
Postoperative complication | 1 month
  We evaluate the presence of postoperative complication such as anastomotic leakage, anastomotic stricture, pneumonia etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Sant'Andrea, Rome, Italy, Italy